CLINICAL TRIAL: NCT06624358
Title: Physical Activity in Adolescents With Chronic Kidney Disease
Brief Title: Physical Activity in CKD
Acronym: PACKD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 23-020727; 1K23DK134847-01A1 (NIH)
Record Dates: First submitted 2024-10-01; First posted 2024-10-03 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-10

CONDITIONS: Chronic Kidney Diseases
Keywords: chronic kidney disease; CKD
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Intervention Model Description: A computerized random number generated by the Way to Health platform will assign children to 1 of 16 study conditions for a 12-week intervention period. The study conditions differ with respect to: personalized exercise plan(on vs off), step goals (ramp-up vs fixed), financial incentive (on vs off), and personalized feedback (on vs off). Our design includes one constant: all participants need to self-monitor their physical activity by wearing the FitBit to allow for daily capture of moderate to vigourous physical activity and step counts. The intervention period is therefore designed to test the effectiveness of 4 components, each with two levels, using a factorial design.
Who Masked: Care Provider, Investigator
Masking Description: Principal investigator and Clinical Care providers will be masked to intervention. Research Coordinator will not be masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (16):
- Fixed step goal only (Experimental): This intervention designed to test if fixed step goals improve physical activity participation.
  Interventions: Behavioral: Increase Physical Activity
- Fixed step goal with feedback (Experimental): This intervention designed to test if fixed step goals and/or daily feed back improve physical activity participation.
  Interventions: Behavioral: Increase Physical Activity
- Fixed step goal with financial incentives (Experimental): This intervention designed to test if fixed step goals and/or financial incentives improve physical activity participation.
  Interventions: Behavioral: Increase Physical Activity
- Fixed step goal with financial incentive and feedback (Experimental): This intervention designed to test if fixed step goals and/or financial incentives and/or daily feedback improve physical activity participation.
  Interventions: Behavioral: Increase Physical Activity
- Ramped Step goals (Experimental): This intervention designed to test if ramped step goals improve physical activity participation.
  Interventions: Behavioral: Increase Physical Activity
- Ramped step goals with feedback (Experimental): This intervention designed to test if ramped step goals and/or daily feedback improve physical activity participation.
  Interventions: Behavioral: Increase Physical Activity
- Ramped step goal with financial incentive (Experimental): This intervention designed to test if ramped step goals and/or financial incentive improve physical activity participation.
  Interventions: Behavioral: Increase Physical Activity
- Ramped step goal with financial incentive and feedback (Experimental): This intervention designed to test if ramped step goals and/or financial incentive and/or daily feedback improve physical activity participation.
  Interventions: Behavioral: Increase Physical Activity
- Personalized plan with fixed step goal (Experimental): This intervention designed to test if personalized exercise plan and/or fixed step goal improves physical activity participation.
  Interventions: Behavioral: Increase Physical Activity
- Personalized plan with fixed step goal and feedback (Experimental): This intervention designed to test if personalized exercise plan and/or fixed step goal and/or daily feedback improves physical activity participation.
  Interventions: Behavioral: Increase Physical Activity
- Personalized plan with fixed step goal and financial incentive (Experimental): This intervention designed to test if personalized exercise plan and/or fixed step goal and/or financial incentive improves physical activity participation.
  Interventions: Behavioral: Increase Physical Activity
- Personalized plan with fixed step goal and financial incentive and feedback (Experimental): This intervention designed to test if personalized exercise plan and/or fixed step goal and/or financial incentive and/or daily feedback improves physical activity participation.
  Interventions: Behavioral: Increase Physical Activity
- Personalized plan with ramped step goal (Experimental): This intervention designed to test if personalized exercise plan and/or fixed step goal improves physical activity participation.
  Interventions: Behavioral: Increase Physical Activity
- Personalized plan with ramped step goal and feedback (Experimental): This intervention designed to test if personalized exercise plan and/or fixed step goal and/or daily feedback improves physical activity participation.
  Interventions: Behavioral: Increase Physical Activity
- Personalized plan with ramped step goal and financial incentive (Experimental): This intervention designed to test if personalized exercise plan and/or fixed step goal and/or financial incentive improves physical activity participation.
  Interventions: Behavioral: Increase Physical Activity
- Personalized plan with ramped step goal and financial incentive and feedback (Experimental): This intervention designed to test if personalized exercise plan and/or fixed step goal and/or financial incentive and/or daily feedback improves physical activity participation.
  Interventions: Behavioral: Increase Physical Activity

INTERVENTIONS:
Behavioral: Increase Physical Activity — Behavioral interventions to improve physical activity

SUMMARY:
The goal of this is to test the efficacy of a 12-week physical activity intervention in 64 adolescents with CKD.

DETAILED DESCRIPTION:
For youth with chronic kidney disease (CKD), cardiovascular disease (CVD) is a leading cause of morbidity and early mortality. Physical activity is a well-recognized determinant of health and quality of life, but, youth with CKD are less physically active than their healthy peers. Identification of effective strategies to increase physical activity in youth with CKD is paramount to improving outcomes. The investigators will test the efficacy of a 12-week physical activity intervention in 64 adolescents with CKD. Guided by the Multiphase Optimization Strategy (MOST) framework, an optimization trial will identify intervention components that increase average daily moderate to vigorous physical activity by 15 min/day, a clinically meaningful increase. The components will be grounded in established behavioral change theories and be delivered via Way to Health, a web-based platform, to overcome barriers at the point of clinical care where time and resources are limited.

ELIGIBILITY:
Inclusion criteria:

For adolescent participants:

1. Males or females age 13 - 18 years
2. Diagnosis of CKD stage II - V not yet on dialysis or with a transplant
3. English proficiency
4. Parental/guardian permission (informed consent), and if applicable, child assent

For caregiver participants:

1. Parent/legal guardian of an enrolled adolescent participant
2. English proficiency

Exclusion Criteria:

For adolescent participants:

1. Pregnant or lactating
2. Non-ambulatory
3. Have high physical activity at baseline (>45 min/day of MVPA)
4. Provide <2 days of physical activity data during the run-in period
5. Have a condition, such as heart or lung disease, that preclude safely engaging in physical activity
6. Have received a solid organ transplant
7. Have limited English proficiency
8. Are on dialysis
9. In the opinion of the investigator, are unable to comply with the requirements of the study protocol or are unsuitable for the study for any reason

For caregivers participants:

1. Limited English proficiency

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-09-30 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Change in time spent in moderate to vigorous physical activity (minutes/day) | pre 12 week intervention and post 12 week intervention
  Change in time spent in moderate to vigorous physical activity measured by Fitbit over the course of 12 weeks

SECONDARY OUTCOMES:
Participant feedback | at the end of the 12 week intervention
  At completion of 12 week intervention, participants will complete an exit survey to collect feedback about the participant's experience. This is not scored.
moderate to vigorous physical activity at 6 months | 6 months
  measure moderate to vigorous physical activity by Fitbit 3 months after completion of 12 week intervention
PROMIS Anxiety | pre 12 week intervention and post 12 week intervention
  Patient self-report of 15 items from PROMIS anxiety domain. Participants rate their experience using a five point scale ranging from never to almost always. Answers are converted to a t-score to compare to the general population. A higher PROMIS T-score represents more of the concept being measured.
PROMIS Depressive Symptoms | pre 12 week intervention and post 12 week intervention
  Patient self-report of 14 items from PROMIS anxiety domain. Participants rate their experience using a five point scale ranging from never to almost always. Answers are converted to a t-score to compare to the general population. A higher PROMIS T-score represents more of the concept being measured.
PROMIS Positive Affect | pre 12 week intervention and post 12 week intervention
  Patient self-report of 39 items from PROMIS positive affect domain. Participants rate their experience using a five point scale ranging from never to always. Answers are converted to a t-score to compare to the general population. A higher PROMIS T-score represents more of the concept being measured.
PROMIS Anger | pre 12 week intervention and post 12 week intervention
  Patient self-report of 9 items from PROMIS anger domain. Participants rate their experience using a five point scale ranging from never to almost always. Answers are converted to a t-score to compare to the general population. A higher PROMIS T-score represents more of the concept being measured.
PROMIS Psychological Stress Experiences | pre 12 week intervention and post 12 week intervention
  Patient self-report of 19 items from PROMIS stress domain. Participants rate their experience using a five point scale ranging from never to always. Answers are converted to a t-score to compare to the general population. A higher PROMIS T-score represents more of the concept being measured.
Change in hand grip strength (age and sex based z-scores) | pre 12-week intervention and post 12-week intervention
  Change in hand grip strength measured by digital hand dynamometer as a age and sex z-score generated from normative data. Z-score is a statistical measurement that describes a values relationship to the mean of a group of values. Values above the mean have positive standard scores, while those below the mean have negative standard scores.
PROMIS Fatigue | pre 12 week intervention and post 12 week intervention
  Patient self-report of 25 items from PROMIS fatigue domain. Participants rate their experience using a five point scale ranging from never to almost always. Answers are converted to a t-score to compare to the general population. A higher PROMIS T-score represents more of the concept being measured.
PROMIS Sleep Disturbance | pre 12 week intervention and post 12 week intervention
  Patient self-report of 15 items from PROMIS sleep disturbance domain. Participants rate their experience using a five point scale ranging from never to almost always. Answers are converted to a t-score to compare to the general population. A higher PROMIS T-score represents more of the concept being measured.
PROMIS Sleep-Related Impairment | pre 12 week intervention and post 12 week intervention
  Patient self-report of 13 items from PROMIS sleep-related impairment domain. Participants rate their experience using a five point scale ranging from never to almost always. Answers are converted to a t-score to compare to the general population. A higher PROMIS T-score represents more of the concept being measured.
PROMIS Life Satisfaction | pre 12 week intervention and post 12 week intervention
  Patient self-report of 42 items from PROMIS life satisfaction domain. Participants rate their experience using a five point scale ranging from never to almost always. Answers are converted to a t-score to compare to the general population. A higher PROMIS T-score represents more of the concept being measured.

CONTACTS AND LOCATIONS:
Overall Officials: Amy Kogon, MD MPH, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
All demographic (without PHI), summary data from clinical tests, survey data, processed summary of physical activity, and summary data from the participant feedback will be shared. The investigators will provide the approved Institutional Review Board (IRB) study protocol and the Management Operating Procedures (MOPs). The sample case report forms and surveys used in the study will be made available. The data dictionary for the project will also be shared. The software versions used in the collection and processing of data will be preserved. Source codes in STATA format used to process data for data cleaning purposes will be preserved and made available.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: Shared data generated from this project will be made available as soon as possible, and no later than the time of publication or the end of the funding period, whichever comes first. The duration of preservation and sharing of the data will be a minimum of 10 years after the end of the funding period.
Access Criteria: Data shall be made available to authorized Arcus users without access restrictions.

REFERENCES:
- [Background] Mitchell JA, Dowda M, Pate RR, Kordas K, Froberg K, Sardinha LB, Kolle E, Page A. Physical Activity and Pediatric Obesity: A Quantile Regression Analysis. Med Sci Sports Exerc. 2017 Mar;49(3):466-473. doi: 10.1249/MSS.0000000000001129. PMID 27755284
- [Background] Clark SL, Denburg MR, Furth SL. Physical activity and screen time in adolescents in the chronic kidney disease in children (CKiD) cohort. Pediatr Nephrol. 2016 May;31(5):801-8. doi: 10.1007/s00467-015-3287-z. Epub 2015 Dec 18. PMID 26684326
- [Background] Fedele DA, Cushing CC, Fritz A, Amaro CM, Ortega A. Mobile Health Interventions for Improving Health Outcomes in Youth: A Meta-analysis. JAMA Pediatr. 2017 May 1;171(5):461-469. doi: 10.1001/jamapediatrics.2017.0042. PMID 28319239
- [Background] Rose T, Barker M, Maria Jacob C, Morrison L, Lawrence W, Strommer S, Vogel C, Woods-Townsend K, Farrell D, Inskip H, Baird J. A Systematic Review of Digital Interventions for Improving the Diet and Physical Activity Behaviors of Adolescents. J Adolesc Health. 2017 Dec;61(6):669-677. doi: 10.1016/j.jadohealth.2017.05.024. Epub 2017 Aug 16. PMID 28822682
- [Background] Groothoff JW, Gruppen MP, Offringa M, Hutten J, Lilien MR, Van De Kar NJ, Wolff ED, Davin JC, Heymans HS. Mortality and causes of death of end-stage renal disease in children: a Dutch cohort study. Kidney Int. 2002 Feb;61(2):621-9. doi: 10.1046/j.1523-1755.2002.00156.x. PMID 11849405
- [Background] McDonald SP, Craig JC; Australian and New Zealand Paediatric Nephrology Association. Long-term survival of children with end-stage renal disease. N Engl J Med. 2004 Jun 24;350(26):2654-62. doi: 10.1056/NEJMoa031643. PMID 15215481
- [Background] Mitsnefes MM, Laskin BL, Dahhou M, Zhang X, Foster BJ. Mortality risk among children initially treated with dialysis for end-stage kidney disease, 1990-2010. JAMA. 2013 May 8;309(18):1921-9. doi: 10.1001/jama.2013.4208. PMID 23645144
- [Background] Laskin BL, Mitsnefes MM, Dahhou M, Zhang X, Foster BJ. The mortality risk with graft function has decreased among children receiving a first kidney transplant in the United States. Kidney Int. 2015 Mar;87(3):575-83. doi: 10.1038/ki.2014.342. Epub 2014 Oct 15. PMID 25317931
- [Background] Parekh RS, Carroll CE, Wolfe RA, Port FK. Cardiovascular mortality in children and young adults with end-stage kidney disease. J Pediatr. 2002 Aug;141(2):191-7. doi: 10.1067/mpd.2002.125910. PMID 12183713
- [Background] Brady TM, Townsend K, Schneider MF, Cox C, Kimball T, Madueme P, Warady B, Furth S, Mitsnefes M. Cystatin C and Cardiac Measures in Children and Adolescents With CKD. Am J Kidney Dis. 2017 Feb;69(2):247-256. doi: 10.1053/j.ajkd.2016.08.036. Epub 2016 Nov 14. PMID 27856090
- [Background] Lalan S, Jiang S, Ng DK, Kupferman F, Warady BA, Furth S, Mitsnefes MM. Cardiometabolic Risk Factors, Metabolic Syndrome, and Chronic Kidney Disease Progression in Children. J Pediatr. 2018 Nov;202:163-170. doi: 10.1016/j.jpeds.2018.06.007. Epub 2018 Jul 2. PMID 30041938
- [Background] Brady TM, Schneider MF, Flynn JT, Cox C, Samuels J, Saland J, White CT, Furth S, Warady BA, Mitsnefes M. Carotid intima-media thickness in children with CKD: results from the CKiD study. Clin J Am Soc Nephrol. 2012 Dec;7(12):1930-7. doi: 10.2215/CJN.03130312. Epub 2012 Sep 13. PMID 22977209
- [Background] Mitsnefes M, Flynn J, Cohn S, Samuels J, Blydt-Hansen T, Saland J, Kimball T, Furth S, Warady B; CKiD Study Group. Masked hypertension associates with left ventricular hypertrophy in children with CKD. J Am Soc Nephrol. 2010 Jan;21(1):137-44. doi: 10.1681/ASN.2009060609. Epub 2009 Nov 16. PMID 19917781
- [Background] Khandelwal P, Murugan V, Hari S, Lakshmy R, Sinha A, Hari P, Bagga A. Dyslipidemia, carotid intima-media thickness and endothelial dysfunction in children with chronic kidney disease. Pediatr Nephrol. 2016 Aug;31(8):1313-20. doi: 10.1007/s00467-016-3350-4. Epub 2016 Feb 26. PMID 26921213
- [Background] Lai HL, Kartal J, Mitsnefes M. Hyperinsulinemia in pediatric patients with chronic kidney disease: the role of tumor necrosis factor-alpha. Pediatr Nephrol. 2007 Oct;22(10):1751-6. doi: 10.1007/s00467-007-0533-z. Epub 2007 Jun 1. PMID 17541791
- [Background] Hooper SR, Johnson RJ, Gerson AC, Lande MB, Shinnar S, Harshman LA, Kogon AJ, Matheson M, Bartosh S, Carlson J, Warady BA, Furth SL. Overview of the findings and advances in the neurocognitive and psychosocial functioning of mild to moderate pediatric CKD: perspectives from the Chronic Kidney Disease in Children (CKiD) cohort study. Pediatr Nephrol. 2022 Apr;37(4):765-775. doi: 10.1007/s00467-021-05158-w. Epub 2021 Jun 10. PMID 34110493
- [Background] Brand C, Martins CML, Lemes VB, Pessoa MLF, Dias AF, Cadore EL, Mota J, Gaya ACA, Gaya AR. Effects and prevalence of responders after a multicomponent intervention on cardiometabolic risk factors in children and adolescents with overweight/obesity: Action for health study. J Sports Sci. 2020 Mar;38(6):682-691. doi: 10.1080/02640414.2020.1725384. Epub 2020 Feb 12. PMID 32050850
- [Background] Savoye M, Caprio S, Dziura J, Camp A, Germain G, Summers C, Li F, Shaw M, Nowicka P, Kursawe R, Depourcq F, Kim G, Tamborlane WV. Reversal of early abnormalities in glucose metabolism in obese youth: results of an intensive lifestyle randomized controlled trial. Diabetes Care. 2014 Feb;37(2):317-24. doi: 10.2337/dc13-1571. Epub 2013 Sep 23. PMID 24062325
- [Background] Herbst A, Kapellen T, Schober E, Graf C, Meissner T, Holl RW; DPV-Science-Initiative. Impact of regular physical activity on blood glucose control and cardiovascular risk factors in adolescents with type 2 diabetes mellitus--a multicenter study of 578 patients from 225 centres. Pediatr Diabetes. 2015 May;16(3):204-10. doi: 10.1111/pedi.12144. Epub 2014 Jun 2. PMID 24888254
- [Background] Brown HE, Pearson N, Braithwaite RE, Brown WJ, Biddle SJ. Physical activity interventions and depression in children and adolescents : a systematic review and meta-analysis. Sports Med. 2013 Mar;43(3):195-206. doi: 10.1007/s40279-012-0015-8. PMID 23329611
- [Background] Elvsaas IKO, Giske L, Fure B, Juvet LK. Multicomponent Lifestyle Interventions for Treating Overweight and Obesity in Children and Adolescents: A Systematic Review and Meta-Analyses. J Obes. 2017;2017:5021902. doi: 10.1155/2017/5021902. Epub 2017 Dec 17. PMID 29391949
- [Background] Jones HM, Al-Khudairy L, Melendez-Torres GJ, Oyebode O. Viewpoints of adolescents with overweight and obesity attending lifestyle obesity treatment interventions: a qualitative systematic review. Obes Rev. 2019 Jan;20(1):156-169. doi: 10.1111/obr.12771. Epub 2018 Oct 29. PMID 30375160
- [Background] Patel MS, Asch DA, Rosin R, Small DS, Bellamy SL, Heuer J, Sproat S, Hyson C, Haff N, Lee SM, Wesby L, Hoffer K, Shuttleworth D, Taylor DH, Hilbert V, Zhu J, Yang L, Wang X, Volpp KG. Framing Financial Incentives to Increase Physical Activity Among Overweight and Obese Adults: A Randomized, Controlled Trial. Ann Intern Med. 2016 Mar 15;164(6):385-94. doi: 10.7326/M15-1635. Epub 2016 Feb 16. PMID 26881417
- [Background] Lappan L, Yeh M-C, Leung MM (2015) Technology as a Platform for Improving Healthy Behaviors and Weight Status in Children and Adolescents: A Review. Obes Open Access 1(3): http://dx.doi. org/10.16966/2380-5528.109
- [Background] Webb TL, Joseph J, Yardley L, Michie S. Using the internet to promote health behavior change: a systematic review and meta-analysis of the impact of theoretical basis, use of behavior change techniques, and mode of delivery on efficacy. J Med Internet Res. 2010 Feb 17;12(1):e4. doi: 10.2196/jmir.1376. PMID 20164043
- [Background] Ajzen, I. (1991). The theory of planned behavior. Organizational Behavior and Human Decision Processes, 50(2), 179-211. https://doi.org/10.1016/0749-5978(91)90020-T
- [Background] Bandura A. Social Learning Theory. Englewood Cliffs, NJ: Prentice Hall; 1977
- [Background] Rice T. The behavioral economics of health and health care. Annu Rev Public Health. 2013;34:431-47. doi: 10.1146/annurev-publhealth-031912-114353. Epub 2013 Jan 7. PMID 23297657
- [Background] Vlaev I, King D, Darzi A, Dolan P. Changing health behaviors using financial incentives: a review from behavioral economics. BMC Public Health. 2019 Aug 7;19(1):1059. doi: 10.1186/s12889-019-7407-8. PMID 31391010
- [Background] Oliver A. Nudges, shoves and budges: Behavioural economic policy frameworks. Int J Health Plann Manage. 2018 Jan;33(1):272-275. doi: 10.1002/hpm.2419. Epub 2017 May 19. PMID 28523778
- [Background] Agarwal A, Patel M. Prescribing Behavior Change: Opportunities and Challenges for Clinicians to Embrace Digital and Mobile Health. JMIR Mhealth Uhealth. 2020 Aug 4;8(8):e17281. doi: 10.2196/17281. PMID 32749997
- [Background] Patel MS, Small DS, Harrison JD, Fortunato MP, Oon AL, Rareshide CAL, Reh G, Szwartz G, Guszcza J, Steier D, Kalra P, Hilbert V. Effectiveness of Behaviorally Designed Gamification Interventions With Social Incentives for Increasing Physical Activity Among Overweight and Obese Adults Across the United States: The STEP UP Randomized Clinical Trial. JAMA Intern Med. 2019 Dec 1;179(12):1624-1632. doi: 10.1001/jamainternmed.2019.3505. PMID 31498375
- [Background] Piper ME, Fiore MC, Smith SS, Fraser D, Bolt DM, Collins LM, Mermelstein R, Schlam TR, Cook JW, Jorenby DE, Loh WY, Baker TB. Identifying effective intervention components for smoking cessation: a factorial screening experiment. Addiction. 2016 Jan;111(1):129-41. doi: 10.1111/add.13162. Epub 2015 Nov 19. PMID 26582269
- [Background] Bernstein SL, Dziura J, Weiss J, Miller T, Vickerman KA, Grau LE, Pantalon MV, Abroms L, Collins LM, Toll B. Tobacco dependence treatment in the emergency department: A randomized trial using the Multiphase Optimization Strategy. Contemp Clin Trials. 2018 Mar;66:1-8. doi: 10.1016/j.cct.2017.12.016. Epub 2017 Dec 27. PMID 29287665
- [Background] Piper ME, Cook JW, Schlam TR, Jorenby DE, Smith SS, Collins LM, Mermelstein R, Fraser D, Fiore MC, Baker TB. A Randomized Controlled Trial of an Optimized Smoking Treatment Delivered in Primary Care. Ann Behav Med. 2018 Sep 13;52(10):854-864. doi: 10.1093/abm/kax059. PMID 30212849
- [Background] Engle JL, Mermelstein R, Baker TB, Smith SS, Schlam TR, Piper ME, Jorenby DE, Collins LM, Cook JW. Effects of motivation phase intervention components on quit attempts in smokers unwilling to quit: A factorial experiment. Drug Alcohol Depend. 2019 Apr 1;197:149-157. doi: 10.1016/j.drugalcdep.2019.01.011. Epub 2019 Feb 16. PMID 30825795
- [Background] Celano CM, Albanese AM, Millstein RA, Mastromauro CA, Chung WJ, Campbell KA, Legler SR, Park ER, Healy BC, Collins LM, Januzzi JL, Huffman JC. Optimizing a Positive Psychology Intervention to Promote Health Behaviors After an Acute Coronary Syndrome: The Positive Emotions After Acute Coronary Events III (PEACE-III) Randomized Factorial Trial. Psychosom Med. 2018 Jul/Aug;80(6):526-534. doi: 10.1097/PSY.0000000000000584. PMID 29624523
- [Background] Phillips SM, Penedo FJ, Collins LM, Solk P, Siddique J, Song J, Cella D, Courneya KS, Ackermann RT, Welch WA, Auster-Gussman LA, Whitaker M, Cullather E, Izenman E, Spring B. Optimization of a technology-supported physical activity promotion intervention for breast cancer survivors: Results from Fit2Thrive. Cancer. 2022 Mar 1;128(5):1122-1132. doi: 10.1002/cncr.34012. Epub 2021 Nov 23. PMID 34812521
- [Background] Pellegrini CA, Hoffman SA, Collins LM, Spring B. Optimization of remotely delivered intensive lifestyle treatment for obesity using the Multiphase Optimization Strategy: Opt-IN study protocol. Contemp Clin Trials. 2014 Jul;38(2):251-9. doi: 10.1016/j.cct.2014.05.007. Epub 2014 May 17. PMID 24846621
- [Background] Spring B, Pfammatter AF, Marchese SH, Stump T, Pellegrini C, McFadden HG, Hedeker D, Siddique J, Jordan N, Collins LM. A Factorial Experiment to Optimize Remotely Delivered Behavioral Treatment for Obesity: Results of the Opt-IN Study. Obesity (Silver Spring). 2020 Sep;28(9):1652-1662. doi: 10.1002/oby.22915. Epub 2020 Jul 12. PMID 32656994
- [Background] Collins LM, Dziak JJ, Kugler KC, Trail JB. Factorial experiments: efficient tools for evaluation of intervention components. Am J Prev Med. 2014 Oct;47(4):498-504. doi: 10.1016/j.amepre.2014.06.021. Epub 2014 Aug 1. PMID 25092122
- [Background] Isoyama N, Qureshi AR, Avesani CM, Lindholm B, Barany P, Heimburger O, Cederholm T, Stenvinkel P, Carrero JJ. Comparative associations of muscle mass and muscle strength with mortality in dialysis patients. Clin J Am Soc Nephrol. 2014 Oct 7;9(10):1720-8. doi: 10.2215/CJN.10261013. Epub 2014 Jul 29. PMID 25074839
- [Background] Kuki A, Tanaka K, Kushiyama A, Tanaka Y, Motonishi S, Sugano Y, Furuya T, Ozawa T. Association of gait speed and grip strength with risk of cardiovascular events in patients on haemodialysis: a prospective study. BMC Nephrol. 2019 May 30;20(1):196. doi: 10.1186/s12882-019-1370-6. PMID 31146702
- [Background] Celis-Morales CA, Welsh P, Lyall DM, Steell L, Petermann F, Anderson J, Iliodromiti S, Sillars A, Graham N, Mackay DF, Pell JP, Gill JMR, Sattar N, Gray SR. Associations of grip strength with cardiovascular, respiratory, and cancer outcomes and all cause mortality: prospective cohort study of half a million UK Biobank participants. BMJ. 2018 May 8;361:k1651. doi: 10.1136/bmj.k1651. PMID 29739772
- [Background] Ho FKW, Celis-Morales CA, Petermann-Rocha F, Sillars A, Welsh P, Welsh C, Anderson J, Lyall DM, Mackay DF, Sattar N, Gill JMR, Pell JP, Gray SR. The association of grip strength with health outcomes does not differ if grip strength is used in absolute or relative terms: a prospective cohort study. Age Ageing. 2019 Sep 1;48(5):684-691. doi: 10.1093/ageing/afz068. PMID 31204772
- [Background] Jang SK, Kim JH, Lee Y. Effect of relative handgrip strength on cardiovascular disease among Korean adults aged 45 years and older: Results from the Korean Longitudinal Study of Aging (2006-2016). Arch Gerontol Geriatr. 2020 Jan-Feb;86:103937. doi: 10.1016/j.archger.2019.103937. Epub 2019 Sep 11. PMID 31574451
- [Background] Leong DP, Teo KK, Rangarajan S, Lopez-Jaramillo P, Avezum A Jr, Orlandini A, Seron P, Ahmed SH, Rosengren A, Kelishadi R, Rahman O, Swaminathan S, Iqbal R, Gupta R, Lear SA, Oguz A, Yusoff K, Zatonska K, Chifamba J, Igumbor E, Mohan V, Anjana RM, Gu H, Li W, Yusuf S; Prospective Urban Rural Epidemiology (PURE) Study investigators. Prognostic value of grip strength: findings from the Prospective Urban Rural Epidemiology (PURE) study. Lancet. 2015 Jul 18;386(9990):266-73. doi: 10.1016/S0140-6736(14)62000-6. Epub 2015 May 13. PMID 25982160
- [Background] Cohen DD, Gomez-Arbelaez D, Camacho PA, Pinzon S, Hormiga C, Trejos-Suarez J, Duperly J, Lopez-Jaramillo P. Low muscle strength is associated with metabolic risk factors in Colombian children: the ACFIES study. PLoS One. 2014 Apr 8;9(4):e93150. doi: 10.1371/journal.pone.0093150. eCollection 2014. PMID 24714401
- [Background] Zhang R, Li C, Liu T, Zheng L, Li S. Handgrip Strength and Blood Pressure in Children and Adolescents: Evidence From NHANES 2011 to 2014. Am J Hypertens. 2018 Jun 11;31(7):792-796. doi: 10.1093/ajh/hpy032. PMID 29529209
- [Background] Rioux BV, Kuwornu P, Sharma A, Tremblay MS, McGavock JM, Senechal M. Association Between Handgrip Muscle Strength and Cardiometabolic z-Score in Children 6 to 19 Years of Age: Results from the Canadian Health Measures Survey. Metab Syndr Relat Disord. 2017 Sep;15(7):379-384. doi: 10.1089/met.2016.0147. Epub 2017 Jul 31. PMID 28759349
- [Background] Foster BJ, Kalkwarf HJ, Shults J, Zemel BS, Wetzsteon RJ, Thayu M, Foerster DL, Leonard MB. Association of chronic kidney disease with muscle deficits in children. J Am Soc Nephrol. 2011 Feb;22(2):377-86. doi: 10.1681/ASN.2010060603. Epub 2010 Nov 29. PMID 21115614
- [Background] Lee DY, Wetzsteon RJ, Zemel BS, Shults J, Organ JM, Foster BJ, Herskovitz RM, Foerster DL, Leonard MB. Muscle torque relative to cross-sectional area and the functional muscle-bone unit in children and adolescents with chronic disease. J Bone Miner Res. 2015 Mar;30(3):575-83. doi: 10.1002/jbmr.2375. PMID 25264231
- [Background] Wind AE, Takken T, Helders PJ, Engelbert RH. Is grip strength a predictor for total muscle strength in healthy children, adolescents, and young adults? Eur J Pediatr. 2010 Mar;169(3):281-7. doi: 10.1007/s00431-009-1010-4. Epub 2009 Jun 14. PMID 19526369
- [Background] Adams MA, Caparosa S, Thompson S, Norman GJ. Translating physical activity recommendations for overweight adolescents to steps per day. Am J Prev Med. 2009 Aug;37(2):137-40. doi: 10.1016/j.amepre.2009.03.016. Epub 2009 Jun 12. PMID 19524391
- [Background] Adams MA, Johnson WD, Tudor-Locke C. Steps/day translation of the moderate-to-vigorous physical activity guideline for children and adolescents. Int J Behav Nutr Phys Act. 2013 Apr 21;10:49. doi: 10.1186/1479-5868-10-49. PMID 23601369
- [Background] Volpp KG, John LK, Troxel AB, Norton L, Fassbender J, Loewenstein G. Financial incentive-based approaches for weight loss: a randomized trial. JAMA. 2008 Dec 10;300(22):2631-7. doi: 10.1001/jama.2008.804. PMID 19066383
- [Background] Wong CA, Miller VA, Murphy K, Small D, Ford CA, Willi SM, Feingold J, Morris A, Ha YP, Zhu J, Wang W, Patel MS. Effect of Financial Incentives on Glucose Monitoring Adherence and Glycemic Control Among Adolescents and Young Adults With Type 1 Diabetes: A Randomized Clinical Trial. JAMA Pediatr. 2017 Dec 1;171(12):1176-1183. doi: 10.1001/jamapediatrics.2017.3233. PMID 29059263
- [Background] Godino JG, Wing D, de Zambotti M, Baker FC, Bagot K, Inkelis S, Pautz C, Higgins M, Nichols J, Brumback T, Chevance G, Colrain IM, Patrick K, Tapert SF. Performance of a commercial multi-sensor wearable (Fitbit Charge HR) in measuring physical activity and sleep in healthy children. PLoS One. 2020 Sep 4;15(9):e0237719. doi: 10.1371/journal.pone.0237719. eCollection 2020. PMID 32886714
- [Background] Latorre Roman PA, Lopez DM, Aguayo BB, Fuentes AR, Garcia-Pinillos F, Redondo MM. Handgrip strength is associated with anthropometrics variables and sex in preschool children: A cross sectional study providing reference values. Phys Ther Sport. 2017 Jul;26:1-6. doi: 10.1016/j.ptsp.2017.04.002. Epub 2017 Apr 5. PMID 28499192
- [Background] Le T, Shim AL, Newman D. Does a relationship between handgrip strength and coincidence anticipation timing exist among young adults: a pilot study. Int J Occup Saf Ergon. 2022 Dec;28(4):2546-2550. doi: 10.1080/10803548.2021.2010377. Epub 2021 Dec 24. PMID 34823437
- [Background] Rajput R, Garg R, Rajput M, Rani M, Darshan An V. Body composition and handgrip strength in patients with prediabetes: A case-control study from Haryana, North India. Diabetes Metab Syndr. 2021 May-Jun;15(3):823-827. doi: 10.1016/j.dsx.2021.03.036. Epub 2021 Apr 9. PMID 33865056
- [Background] Pereira RA, Cordeiro AC, Avesani CM, Carrero JJ, Lindholm B, Amparo FC, Amodeo C, Cuppari L, Kamimura MA. Sarcopenia in chronic kidney disease on conservative therapy: prevalence and association with mortality. Nephrol Dial Transplant. 2015 Oct;30(10):1718-25. doi: 10.1093/ndt/gfv133. Epub 2015 May 21. PMID 25999376
- [Background] Carrero JJ, Chmielewski M, Axelsson J, Snaedal S, Heimburger O, Barany P, Suliman ME, Lindholm B, Stenvinkel P, Qureshi AR. Muscle atrophy, inflammation and clinical outcome in incident and prevalent dialysis patients. Clin Nutr. 2008 Aug;27(4):557-64. doi: 10.1016/j.clnu.2008.04.007. Epub 2008 Jun 6. PMID 18538898
- [Background] Matsuzawa R, Matsunaga A, Wang G, Kutsuna T, Ishii A, Abe Y, Takagi Y, Yoshida A, Takahira N. Habitual physical activity measured by accelerometer and survival in maintenance hemodialysis patients. Clin J Am Soc Nephrol. 2012 Dec;7(12):2010-6. doi: 10.2215/CJN.03660412. Epub 2012 Sep 13. PMID 22977216
- [Background] Robinson-Cohen C, Littman AJ, Duncan GE, Weiss NS, Sachs MC, Ruzinski J, Kundzins J, Rock D, de Boer IH, Ikizler TA, Himmelfarb J, Kestenbaum BR. Physical activity and change in estimated GFR among persons with CKD. J Am Soc Nephrol. 2014 Feb;25(2):399-406. doi: 10.1681/ASN.2013040392. Epub 2013 Dec 12. PMID 24335971
- [Background] Hogan J, Schneider MF, Pai R, Denburg MR, Kogon A, Brooks ER, Kaskel FJ, Reidy KJ, Saland JM, Warady BA, Furth SL, Patzer RE, Greenbaum LA. Grip strength in children with chronic kidney disease. Pediatr Nephrol. 2020 May;35(5):891-899. doi: 10.1007/s00467-019-04461-x. Epub 2020 Jan 13. PMID 31932960
- [Background] Brener ND, Kann L, McManus T, Kinchen SA, Sundberg EC, Ross JG. Reliability of the 1999 youth risk behavior survey questionnaire. J Adolesc Health. 2002 Oct;31(4):336-42. doi: 10.1016/s1054-139x(02)00339-7. PMID 12359379
- [Background] Sekhon M, Cartwright M, Francis JJ. Acceptability of healthcare interventions: an overview of reviews and development of a theoretical framework. BMC Health Serv Res. 2017 Jan 26;17(1):88. doi: 10.1186/s12913-017-2031-8. PMID 28126032
- [Background] NIDDK. NIDDK Strategic Plan for Research (Dec. 2021). Dec 2021. NIH Publication Number: 21-DK-8159. https://www.niddk.nih.gov/about-niddk/strategic-plans-reports/niddk-strategic-plan-for-research. Accessed February 10, 2022.
- [Background] Collins L, Optimization of Behvioral, Biobehavioral and Biomedial Interventions. Springer International Publishing; 2018.
- [Background] Collins L, Huang L DJ. R Package MOST: Multiphase Optimization Strategy. 2017.
- [Background] Troiano RP, Berrigan D, Dodd KW, Masse LC, Tilert T, McDowell M. Physical activity in the United States measured by accelerometer. Med Sci Sports Exerc. 2008 Jan;40(1):181-8. doi: 10.1249/mss.0b013e31815a51b3. PMID 18091006